CLINICAL TRIAL: NCT07407413
Title: The Edu:Social Health Care Project: Investigating the Effects of an Online Socio-emotional Dyad Intervention on Healthcare Students' Mental Health, Resilience, Social Competencies and Behaviors
Brief Title: Online Socio-emotional Dyad Training for Healthcare Students' Well-being and Social Skills
Acronym: EduSocHealth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Social Neuroscience Lab (Other)
Collaborators: Paracelsus Medizinische Privatuniversität (PMU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Edu:Social Health Care Project
Record Dates: First submitted 2026-01-12; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Intervention Condition; Control (Delayed Training) Condition
Keywords: Mental Training; Dyad Training; Compassionate-Listening; Empathic-Listening; Empathy; Compassion; Mental-Health; Online & App-based Training; Resilience; Social Cohesion; Social Kills; AI-based Voice Assessment; Healthcare students
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: After pre-screening and randomized allocation to the two groups, participants and coordination staff need to be aware of which intervention arm (EmCo intervention group or WCG group) the participant belongs to in order to be able to group into appropriate coaching slots and onboarding I and II sessions prior to starting the actual 8-week online interventions with daily Dyad practice. Outcome assessors and investigators remain blinded to participant allocation for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empathy- and compassion-based socio-emotional mental training (EmCo) (Experimental): The socio-emotional intervention will consist of two 1.5h online onboarding I and II sessions and then 8 weeks of weekly 1.5-hour online coaching sessions with expert teachers as well as daily dyad practice with a partner over 8 weeks.
  Interventions: Behavioral: Experimental: Empathy- and compassion-based socio-emotional mental training (EmCo)
- Waitlist Control Group (WCG) (Other): Initially, participants in the waitlist control group will not receive the intervention and will be offered the EmCo training only after the intervention group has completed the EmCo training program.
  Interventions: Other: Waitlist Control Group (WCG)

INTERVENTIONS:
Behavioral: Experimental: Empathy- and compassion-based socio-emotional mental training (EmCo) — 1. Participants engage in a structured 13-minute partner-based contemplative exercise. Each dyad reflects on two experiences from the previous 24 hours: one involving a difficult emotion and one involving gratitude. Partners take turns speaking while the other listens non-judgmentally. During weeks 1-4, the practice emphasizes empathic listening; during weeks 5-8, compassionate listening. Participants are instructed to attend to bodily sensations associated with the emotions described. The practice aims to improve coping with difficult emotions, empathic and compassionate listening, (self)acceptance, compassion, gratitude, resilience.
  2. Participants also attend eight 1.5-hour online group sessions led by Expert Dyad teachers. The coaching sessions help deepen the Dyad practice and educate teachers about body language, coping better with difficult emotions/stress, the benefits of empathy versus compassion and the act of listening from a mindset of empathy versus compassion.
  Arms: Empathy- and compassion-based socio-emotional mental training (EmCo)
Other: Waitlist Control Group (WCG) — Participants in the control group will not receive the intervention. They will complete pre- and post-test procedures consisting primarily of self-report questionnaires, and behavioral tasks, as well as ecological momentary assessment (EMA) conducted on four days within two weeks at pre-test and post-test 1 & 2.
  Arms: Waitlist Control Group (WCG)

SUMMARY:
In this Edu:Social Health Care project, a randomized controlled trial with a socio-emotional intervention and a waitlist control group will be conducted to evaluate the effects of a partner-based empathy-compassion Dyad mental training (EmCo) intervention on healthcare students with regard to the following primary outcome domains: 1) mental health, 2) resilience, 3) social cohesion and support, 4) social skills, 5) coping and emotion regulation, and 6) social behaviors.

One main goal is to examine the effects of such adapted 8-week EmCo Dyad intervention within the health care context, with a particular focus on strengthening students' mental health, resilience, social skills and behaviors, and social cohesion as well as fostering interprofessional attitudes by pairing every week study partners across different healthcare disciplines with each other for practicing their daily Dyads (e.g., nursing students will practice daily via app with medical students).

A further aim is to validate the novel Dyad Voice Assessment (DYVA) task, which explores the use of app-based voice recordings as indicators of students' emotional states during their daily partner-based Dyad practice. By combining students' self-reported practice-related emotions with partner-based evaluations, this approach aims to generate new and innovate, more objective markers of training-induced changes in emotional processing and regulation over time in a real-live applied setting.

The final aim is to investigate the cognitive and affective mechanisms and factors underlying observed changes in students' mental health, resilience, social cohesion, social skills and social behaviors, that may explain observed training-related effects in primary outcome domains. Based on previous research, we expect the socio-emotional EmCo Dyad training to activate evolutionary old care- and affiliation-based motivational systems that foster positive affect and motivation, acceptance, trust social capacities and behavioral tendencies. These processes should go along with reduction in loneliness, stress and other mental vulnerabilities (anxiety, depression, burn-out etc.) and foster social skills such as empathy, compassion as well as social cohesion and resilience.

DETAILED DESCRIPTION:
One-quarter to one-third of university students experience a common mental health disorder each year, with evidence indicating rising distress and declining well-being over time. Healthcare students appear particularly vulnerable, showing increasing levels of burnout associated with poorer academic engagement and impaired professional development. Mindfulness- and compassion-based interventions, as well as socio-emotional learning programs, have shown promise in improving mental health outcomes such as depression, anxiety, stress, and burnout, and in strengthening resilience among healthcare students.

In recent years, classic mindfulness-based interventions focusing on individual mental practices have been expanded to include partner-based social practices, known as Dyads, which particularly target social skills such as empathy, (self-)compassion, and social cohesion. However, despite growing research on student well-being, partner-based Dyadic interventions have not yet been systematically investigated in healthcare student populations. Available evidence suggests that Dyads may be more effective than solitary mindfulness practices in reducing loneliness and social stress, strengthening social connection and cohesion, and enhancing resilience and optimism. Moreover, findings indicate that dyadic social practices engage mechanisms that differ from those underlying traditional mindfulness-based interventions.

Empathy, (self-)compassion, and deep listening are core socio-emotional skills in healthcare, supporting effective communication and emotional understanding. However, empathy can lead to empathic distress when individuals are repeatedly exposed to others' suffering, whereas compassion is considered more protective, as it relies on altruistic and care-based motivational systems associated with positive affect and regulatory processes that buffer emotional overwhelm. Despite this distinction, empathy and compassion have not yet been systematically taught to healthcare students in an evidence-based manner. To address this gap, the Edu:Social Health Care project implements the empathy-compassion Dyad training program (EmCo), which trains students to distinguish between empathy and empathic listening and empathy regulation to avoid moving into empathic distress during the first four weeks, and (self)compassion and compassionate listening during the subsequent four weeks.

The EmCo program builds on the Affect Dyad developed in the ReSource project and the online Dyad coaching format implemented in the CovSocial project, both of which demonstrated the effectiveness of partner-based dyadic mental training in inducing brain plasticity, reducing stress, enhancing psychological resilience, and strengthening social cohesion across multiple indicators of biopsychosocial health. In contrast, to the ReSource and CovSocial projects, the present program, includes a novel empathy versus compassion listening component to it. Further, compared with earlier 10-week online Dyad programs, EmCo reduces the intervention duration to eight weeks, aligning with standard mindfulness-based interventions such as MBSR and MBCT and improving feasibility for implementation in healthcare and educational settings.

Accordingly, the study is implemented as a randomized controlled trial in a sample of healthcare students (target N = 360). A multimethod assessment strategy will be used, including self-report validated trait and state questionnaires, behavioral computer tasks delivered at home through webapp, and ecological momentary assessment (EMA) methods based on push-notifications by the app. These different assessments are capturing changes across mental health, resilience, social cohesion and support, social skills, coping and emotion regulation, and social behaviors (e.g., listening, attachment behaviors).

After providing informed consent, participants will be randomized to one of two groups: (1) an empathy-compassion training group (EmCo), based on the Affect Dyad mental practice, or (2) a waitlist control group (WCG). All participants will first complete the pre-test assessment phase including baseline psychometrics, computer-based tasks, and EMA measures. The intervention group will then be onboarded into the intervention with two Online onboarding I and II sessions lead by professional Dyad teachers and then complete the EmCo training program delivered via a dedicated web and smartphone application with daily partner-based Dyads as well as weekly 1.5 hours online coaching sessions. During this period, participants will complete brief weekly self-report questionnaires, Ecological Momentary Assessments (EMA) and daily pre-post Dyad practice ratings (DPR), to capture changes in key psychological and social processes to be used as mediator variables. At the end of the intervention, all participants will complete a post-test phase similar to the pre-test but with an additional final feedback questionnaire.

Following completion of the initial post-test (T1), participants in the waitlist control group will subsequently receive the same 8-week socio-emotional Dyad intervention (EmCo) and complete an additional post-test assessment (T2).

The study was preregistered on the Open Science Framework (OSF) and is publicly available at https://osf.io/3t8s4.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18- and 65-years old.
2. actively enrolled student at the PMU.
3. Proficient in German.
4. Informed consent.
5. No symptoms of psychiatric disease within the past two years.
6. Stable internet access and necessary technical equipment (computer or laptop or tablet, and mobile phone with internet access).
7. No regular contemplative practice (≤ 50 hours total within the past six months); healthy population, non-clinical population.

   Exclusion Criteria:
8. Insufficient German proficiency.
9. Lack of stable internet access or required devices (computer or laptop or tablet, and mobile phone with internet access).
10. No informed consent.
11. Not actively enrolled at PMU.
12. Regular contemplative practice (> 50 hours in the past six months (e.g., dyad, mindfulness, compassion-based practices).
13. Current psychiatric diagnosis or therapy, or reaching screening cutoffs on:

    * Patient Health Questionnaire-9 (PHQ-9; Martin et al., 2006; Löwe et al., 2004; Cutoff ≥ 10),
    * Generalized Anxiety Disorder-7 (GAD-7; Löwe et al., 2007; Spitzer et al., 2006; Cutoff ≥ 10),
    * Toronto Alexithymia Scale-20 (TAS-20; Bagby et al., 1994; Ritz & Kannapin, 2000; Cutoff ≥ 61)
    * Standardized Assessment of Personality - Abbreviated Scale (SAPAS; Moran et al., 2003; Söchtig et al., 2012, Cutoff ≥ 4).
    * Moreover, participants endorsing suicidality on the PHQ-9 will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring depression, anxiety, and stress (Henry & Crawford, 2005; Nilges & Essau, 2021). Higher scores indicate more depression, anxiety, and stress.
Maslach Burnout Inventory-Students Survey (MBI-SS) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring burnout (Gumz et al., 2013; Maslach & Jackson, 1981). Higher scores indicate more burnout.
UCLA Loneliness Scale (UCLA) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring loneliness severity (Döring & Bortz, 1993; Russell et al., 1980). Higher scores indicate more loneliness.
Connor Davidson Resilience Scale (CD-RISC) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring psychological resilience (Connor & Davidson, 2003; Sarubin et al., 2015). Higher scores indicate more resilience.
Social closeness (IOS per profession) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring the felt closeness between persons or groups/communities using a visual representation (Aron et al., 1992; Kinnunen & Windmann, 2013). Higher score indicates more social closeness.
Interprofessionalism Scale (IPAS-D) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale (Norris et al., 2015; Pedersen et al., 2020) measuring attitudes that relate to the Core Competencies for Interprofessional Collaborative Practice (IPEC Report, 2011). Higher scores indicate more positive attitudes toward collaborative practice.
Social Support Scale (F-SozU K-6) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A scale measuring the subjective feeling of having support available (Kliem et al., 2015). Higher scores indicate greater perceived social support.
Socio-Affective Video Task (SoVT) | Assessed at baseline (pre-test), after 4 weeks of empathic listening training (mid-intervention) and after the 4 weeks of compassionate listening training (post-test 1 & 2)
  This task assesses behavioral empathy and compassion using emotional video clips (Klimecki et al., 2014). Higher scores indicate more empathy or more compassion.
Sussex-Oxford Compassion Scale for Self and Others (SOCS) | Assessed at baseline (pre-test), after 4 weeks of empathic listening training (mid-intervention) and after the 4 weeks of compassionate listening training (post-test 1 & 2)
  A scale measuring self-compassion (SOCS-S) and compassion for others (SOCS-O; Gu et al., 2020). Higher scores indicate more compassion.
Mentalization Scale (MENTS) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2).
  A scale measuring the capacity of envisioning one's and others' behaviors with reference to the underlying mental states (Dimitrijević et al., 2018). Higher scores suggesting a more sophisticated capacity for mentalizing.
Prosodic Features of Vocalized Emotional Expressions | Assessed weekly from week 1 to week 8, as part of the Dyad Voice Assessment (DYVA)
  Acoustic assessment of prosodic speech features during participants' daily Dyad practice, analyzed using audEERING devAIce software. The following parameters will be assessed: pitch (Hz), loudness (unitless), speaking rate (syllables per second), and intonation (unitless).
Affect Dimensions of Vocalized Emotional Expressions | Assessed weekly from week 1 to week 8, as part of the Dyad Voice Assessment (DYVA)
  Assessment of continuous affective dimensions of vocalized emotional expressions during participants' daily Dyad practice using audEERING devAIce software. The following parameters will be assessed: arousal, valence, and dominance (each ranging from -1 to 1). Based on arousal-valence scores, the following affect quadrant values will be calculated: high-arousal-high-valence, low-arousal-high-valence, low-arousal-low-valence, and high-arousal-low-valence.
Affect Categories of Vocalized Emotional Expressions | Assessed weekly from week 1 to week 8, as part of the Dyad Voice Assessment (DYVA)
  Classification of vocalized emotional expressions into affect categories during participants' daily Dyad practice using audEERING devAIce software. The following categories will be assessed: angry, happy, and sad, expressed as unitless values ranging from 0 to 1 representing category likelihood.
Stress intensity | Assessed using an EMA design with five push-notification measurements per day, distributed across five 3-hour intervals, on four days within a two-week period, at pre-test (Baseline) and after the 8-week intervention period (post-intervention).
  Custom items based on the Stress Appraisal Measure (SAM; Delahaye et al., 2015; Peacock & Wong, 1990) measuring stress intensity. Higher scores indicate more intense stress.
Coping strategies | Assessed using an EMA design with five push-notification measurements per day, distributed across five 3-hour intervals, on four days within a two-week period, at pre-test (Baseline) and after the 8-week intervention period (post-intervention).
  Custom items based on the Brief-COPE (Carver, 1997; Knoll et al., 2005) and Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski et al., 2001; Loch et al., 2011) measuring Coping Strategies (Acceptance, Positive Reinterpretation, Social Support, Rumination, Self-Blame, Distraction). Higher scores indicate a higher use of the specified coping strategies.
Active Empathic Listening Scale (AELS) | Assessed at baseline (pre-test), after 4 weeks of empathic listening training (mid-intervention) and after the 4 weeks of compassionate listening training (post-test 1 & 2)
  A scale measuring active empathic listening (Bodie, 2011). Higher scores indicate more active empathic listening.
Attachment behavior (ASQ) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  A self-report questionnaire measuring attachment-related behaviors in interpersonal relationships, including proximity seeking, avoidance, and security (Hexel, 2004). Higher scores indicate more pronounced attachment-related behaviors.

SECONDARY OUTCOMES:
Positive Affect (Affect Grid) (explanatory mechanism) | Assessed weekly during the course of 8 weeks of intervention
  Assessment of emotional state (valence) and arousal (Russell et al., 1989). Higher scores on valence and arousal indicate more positive affect and higher arousal.
Emotion Acceptance (EAQ) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A self-report questionnaire measuring emotional awareness, and acceptance of emotions (Beblo et al., 2011; Kisley et al., 2025). Higher scores indicate greater emotion awareness and acceptance
Gratitude Questionnaire-6 (GQ-5-G) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A scale measuring gratitude (Hudecek et al., 2021; McCullough et al., 2002). Higher scores indicate more gratitude.
Self-Kindness Scale (SCS-SF) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A self-report questionnaire measuring self-kindness and compassionate attitudes toward oneself (Hupfeld & Ruffieux, 2011; Raes et al., 2011). Higher scores indicate greater self-kindness.
Positive Interpretation Bias (ERT) (explanatory mechanism) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  This task assesses the tendency to judge persons' facial expressions more positively using morphed sequences of facial expressions (DeBruine & Jones, 2017; Griffiths et al., 2015). Higher scores indicate a stronger positive interpretation bias.
Mentalizing (MENTS) Scale (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A self-report questionnaire measuring the capacity to understand one's own and others' mental states (Dimitrijević et al., 2018). Higher scores indicate greater mentalizing ability.
Short Loneliness Scale (SLS) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A short scale measuring frequency, intensity, and duration of loneliness (Hughes et al., 2004; Qualter et al., 2021). Higher scores indicate more loneliness.
Perceived Stress (PSS-10) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A self-report questionnaire measuring the degree to which situations in one's life are appraised as stressful (Cohen et al., 1983; Klein et al., 2016). Higher scores indicate greater perceived stress.
Depression (PHQ-2) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A brief self-report screening measure assessing core depressive symptoms, including depressed mood and anhedonia (Kroenke et al., 2003). Higher scores indicate greater depressive symptom severity.
Empathic Concern & Distress (IRI) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A scale measuring different facets of social emotions, including personal distress and empathic concern (Davis, 1980; Paulus, 2009). Higher scores indicate higher personal distress or empathic concern.
Trust (KUSIV3) (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  A self-report questionnaire measuring generalized interpersonal trust, including trust in others' reliability and integrity (Beierlein et al., 2012). Higher scores indicate greater interpersonal trust.
In-group-Out-group bias (ERT) (explanatory mechanism) | Assessed at baseline (pre-test) and after the 8-week intervention period (post-test 1 & 2)
  This task assesses the tendency to judge persons from one's own group to be more positive in facial emotion recognition using morphed sequences of facial expressions (DeBruine & Jones, 2017; Griffiths et al., 2015). Higher scores indicate a stronger in-group-out-group bias.
Coping strategies (explanatory mechanism) | Assessed weekly during the course of 8 weeks
  Custom items based on the Brief-COPE (Carver, 1997; Knoll et al., 2005) and Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski et al., 2001; Loch et al., 2011) measuring Coping Strategies (Acceptance, Positive Reinterpretation, Social Support, Rumination, Self-Blame, Distraction). Higher scores indicate a higher use of the specified coping strategies.
DPR-Affect (Affect Grid; explanatory mechanism) | Assessed for 8 weeks during intervention period, before the daily exercise
  Assessment of emotional state (valence) and arousal (Russell et al., 1989) just before starting the Dyad. Higher scores on valence and arousal indicate more positive affect and higher arousal.
DPR-involvement (explanatory mechanism) | Assessed for 8 weeks during intervention period, only in the intervention group, after the daily exercise
  Assessment of listening involvement (1 custom item; only post-Dyad exercise). Higher scores indicate more listening involvement.
Dyad closeness - Inclusion of Other in Self Scale (explanatory mechanism) | Assessed for 8 weeks during intervention period, only in the intervention group, after the daily exercise
  Assessment of how close participants felt to their Dyad partner (post-Dyad exercise). Higher scores indicate more closeness (Aron et al., 1992; Kinnunen & Windmann, 2013).
Dyad listening quality (DPR- listening-quality) | Assessed weekly from week 1 to week 8, after the Dyad practice
  Custom items (self-generated) measuring the quality of listening to the Dyad partner. Higher scores indicate a higher degree of active, attentive listening
DPR-Emotions | Assessed weekly from week 1 to week 8, as part of the Dyad Voice Assessment (DYVA)
  Emotion intensities (of e.g., happiness, gratitude, sadness, anger) rated by the speaker and by the listener of a Dyad directly after the Dyad.
DPR-Listening-Affect | Assessed weekly from week 1 to week 8, after the Dyad practice
  Custom items (self-generated) measuring the self-rated affective state during listening to the Dyad partner's telling of the difficult situation and the event that they are grateful for. Higher scores indicate a more positive affect.
Dyad empathic and compassionate listening skills (DPR-listening-skills) | Assessed weekly from week 1 to week 8, after the Dyad practice
  Custom items (self-generated) measuring the self-rated skill of listening empathically and compassionately to the Dyad partner's telling of the difficult situation and the event that they are grateful for. Higher scores indicate a higher degree of empathic or compassionate listening respectively.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9; pre-screening) | Assessed before the intervention, only once, to pre-screen out from the study individuals who have clinical levels of depressive symptoms
  A scale assessing depression (Löwe et al., 2004; Martin et al., 2006). Higher scores indicate more depression.
Generalized Anxiety Disorder (GAD-7; pre-screening) | Assessed prior to the intervention, only once, to pre-screen out from the study individuals who have clinical levels of anxious symptoms
  A scale assessing generalized anxiety (Spitzer et al., 2006; Löwe et al., 2007). Higher scores indicate more anxiety.
Toronto Alexithymia Scale (TAS-20; pre-screening) | Assessed before the intervention, only once, to pre-screen out from the study individuals who have high levels of alexithymia
  A scale assessing alexithymia (Bagby et al., 1994; Ritz & Kannapin, 2000). Higher scores indicate more alexithymia.
Standardized Assessment of Personality - Abbreviated Scale (SAPAS; pre-screening) | Assessed before the intervention, only once, to pre-screen out from the study individuals who have high levels of personality disorders symptoms
  A self-report scale used to screen personality disorders (Moran et al., 2003; Söchtig et al., 2012).
General demographic questions | Assessed before the intervention, only once, to collect demographic information
  Self-generated demographic items.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Singer, Ph.D., Principal Investigator — Social Neuroscience Lab, Max Planck Society

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Aron, A., Aron, E. N., & Smollan, D. (1992). Inclusion of Other in the Self Scale and the structure of interpersonal closeness. Journal of Personality and Social Psychology, 63(4), 596-612. https://doi.org/10.1037/0022-3514.63.4.596
- [Background] 2. Auerbach, R. P., Mortier, P., Bruffaerts, R., Alonso, J., Benjet, C., Cuijpers, P., Demyttenaere, K., Ebert, D. D., Green, J. G., Hasking, P., Murray, E., Nock, M. K., Pinder-Amaker, S., Sampson, N. A., Stein, D. J., Vilagut, G., Zaslavsky, A. M., Kessler, R. C., & WHO WMH-ICS Collaborators. (2018). WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. Journal of Abnormal Psychology, 127(7), 623-638. https://doi.org/10.1037/abn0000362
- [Background] 3. Auerbach, R. P., Mortier, P., Bruffaerts, R., Murray, E., & Sampson, N., et al. (2016). Mental disorders among college students in the World Health Organization World Mental Health Surveys. Psychological Medicine, 46(14), 2955-2970. https://doi.org/10.1017/S0033291716001665
- [Background] 4. Bagby, R. M., Parker, J. D., & Taylor, G. J. (1994). The twenty-item Toronto Alexithymia Scale-I. Item selection and cross-validation of the factor structure. Journal of psychosomatic research, 38(1), 23-32. https://doi.org/10.1016/0022-3999(94)90005-1
- [Background] 5. Barbosa, P., Raymond, G., Zlotnick, C., Wilk, J., Toomey III, R., & Mitchell III, J. (2013). Mindfulness-based stress reduction training is associated with greater empathy and reduced anxiety for graduate healthcare students. Education for health, 26(1), 9-14. https://doi.org/10.4103/1357-6283.112794
- [Background] 6. Beblo, T., Scheulen, C., Fernando, S. C., Griepenstroh, J., Aschenbrenner, S., Rodewald, K. & Driessen, M. (2011). Psychometrische Analyse eines neuen Fragebogens zur Erfassung der Akzeptanz von unangenehmen und angenehmen Gefühlen (FrAGe). Zeitschrift Für Psychiatrie, Psychologie Und Psychotherapie, 59(2), 133-144. https://doi.org/10.1024/1661-4747/a000063
- [Background] 7. Beck, R. S., Daughtridge, R., & Sloane, P. D. (2002). Physician-patient communication in the primary care office: a systematic review. The Journal of the American Board of Family Practice, 15(1), 25-38.
- [Background] 8. Beierlein, C., Kemper, C. J., Kovaleva, A., & Rammstedt, B. (2012). Kurzskala zur Messung des zwischenmenschlichen Vertrauens: die Kurzskala Interpersonales Vertrauen (KUSIV3). (GESIS-Working Papers, 2012/22). Mannheim: GESIS - Leibniz-Institut für Sozialwissenschaften. https://nbn-resolving.org/urn:nbn:de:0168-ssoar-312126
- [Background] 9. Bodie, G. D. (2011). The Active-Empathic Listening Scale (AELS): Conceptualization and Evidence of Validity Within the Interpersonal Domain. Communication Quarterly, 59(3), 277-295. https://doi.org/10.1080/01463373.2011.583495
- [Background] 10. Bullock, G., Kraft, L., Amsden, K., Gore, W., Prengle, B., Wimsatt, J., Ledbetter, L., Covington, K., & Goode, A. (2017). The prevalence and effect of burnout on graduate healthcare students. Canadian medical education journal, 8(3), e90-e108. https://journalhosting.ucalgary.ca/index.php/cmej/article/view/36890
- [Background] 11. Carver, C. S. (1997). You want to measure coping but your protocol's too long: Consider the brief cope. International Journal of Behavioral Medicine, 4(1), 92-100. https://doi.org/10.1207/s15327558ijbm0401_6
- [Background] 12. Cohen, S., Kamarck, T., & Mermelstein, R. (1983). Perceived Stress Scale [Database record]. APA PsycTests. https://doi.org/10.1037/t02889-000
- [Background] 13. Connor, K. M., & Davidson, J. R. (2003). Development of a new resilience scale: The Connor-Davidson resilience scale (CD-RISC). Depression and anxiety, 18(2), 76-82. https://doi.org/10.1002/da.10113
- [Background] 14. Curran, T., & Hill, A. P. (2019). Perfectionism is increasing over time: A meta-analysis of birth cohort differences from 1989 to 2016. Psychological Bulletin, 145(4), 410-429. https://doi.org/10.1037/bul0000138
- [Background] 15. Davis, M. H. (1980). A multidimensional approach to individual differences in empathy. JSAS Catalog of Selected Documents in Psychology, 1980, 10, p. 85. https://www.uv.es/friasnav/Davis_1980.pdf
- [Background] 16. DeBruine, L. & Jones, B. (2017). Face Research Lab London Set. figshare. Dataset. https://doi.org/10.6084/m9.figshare.5047666.v5
- [Background] 17. Delahaye, M., Stieglitz, R. D., Graf, M., Keppler, C., Maes, J., & Pflueger, M. (2015). German translation and validation of the stress appraisal measure (SAM). Fortschritte der Neurologie-psychiatrie, 83(5), 276-285. https://doi.org/10.1055/s-0034-1399727
- [Background] 18. Derksen, F., Bensing, J., & Lagro-Janssen, A. (2013). Effectiveness of empathy in general practice: A systematic review. British Journal of General Practice, 63(606), e76-e84. https://doi.org/10.3399/bjgp13X660814
- [Background] 19. Dimitrijević, A., Hanak, N., Altaras Dimitrijević, A., & Jolić Marjanović, Z. (2018). The Mentalization Scale (MentS): A self-report measure for the assessment of mentalizing capacity. Journal of Personality Assessment, 100(3), 268-280. https://doi.org/10.1080/00223891.2017.1310730
- [Background] 20. Döring, N., & Bortz, J. (1993). Psychometrische Einsamkeitsforschung: Deutsche Neukonstruktion der UCLA Loneliness Scale. Diagnostica, 39(3), 224-239.
- [Background] 21. Gandía-Carbonell, N., Molla-Esparza, C., Lorente, S., Viguer, P., & Losilla, J. M. (2025). Strategies to assess and promote the socio-emotional competencies of university students in the socio-educational and healthcare fields: A scoping review. PLoS One, 20(5), e0324531. https://doi.org/10.1371/journal.pone.0324531
- [Background] 22. Garnefski, N., Kraaij, V., & Spinhoven, P. (2001). Negative life events, cognitive emotion regulation and emotional problems. Personality and Individual differences, 30(8), 1311-1327. https://doi.org/10.1016/S0191-8869(00)00113-6
- [Background] 23. Godara, M., Hecht, M., & Singer, T. (2024). Training-related improvements in mental well-being through reduction in negative interpretation bias: A randomized trial of online socio-emotional dyadic and mindfulness interventions. Journal of Affective Disorders, 354, 662-672. https://doi.org/10.1016/j.jad.2024.03.037
- [Background] 24. Godara, M., Silveira, S., Matthäus, H., Heim, C., Voelkle, M., Hecht, M., Binder, E. B., & Singer, T. (2021). Investigating differential effects of socio-emotional and mindfulness-based online interventions on mental health, resilience and social capacities during the COVID-19 pandemic: The study protocol. PLOS ONE, 16(11), e0256323. https://doi.org/10.1371/journal.pone.0256323
- [Background] 25. Godara, M. & Singer, T. (2024a). 10-Week Trajectories of Candidate Psychological Processes Differentially Predict Mental Health Gains from Online Dyadic Versus Mindfulness Interventions: A Randomized Clinical Trial. Journal of Clinical Medicine 13 (11), 3295. https://doi.org/10.3390/jcm13113295
- [Background] 26. Godara, M. & Singer, T. (2024b). Resilient Stress Reactivity Profiles Predict Mental Health Gains from Online Contemplative Training: A Randomized Clinical Trial. Journal of Personalized Medicine 14 (5), 493. https://doi.org/10.3390/jpm14050493
- [Background] 27. Griffiths, S., Jarrold, C., Penton-Voak, I. S., & Munafò, M. R. (2015). Feedback training induces a bias for detecting happiness or fear in facial expressions that generalises to a novel task. Psychiatry Research, 230(3), 951-957. https://doi.org/10.1016/j.psychres.2015.11.007
- [Background] 28. Gu, J., Baer, R., Cavanagh, K., Kuyken, W., & Strauss, C. (2019). Development and psychometric properties of the Sussex-Oxford compassion scales (SOCS). Assessment, 27(1), 3-20. https://doi.org/10.1177/1073191119860911
- [Background] 29. Gumz, A., Erices, R., Brähler, E., & Zenger, M. (2013). Faktorstruktur und Gütekriterien der deutschen Übersetzung des Maslach-Burnout-Inventars für Studierende von Schaufeli et al. (MBI-SS) [Factorial structure and psychometric criteria of the German translation of the Maslach Burnout Inventory-Student Version by Schaufeli et al. (MBI-SS)]. PPmP: Psychotherapie Psychosomatik Medizinische Psychologie, 63(2), 77-84. https://doi.org/10.1055/s-0032-1323695
- [Background] 30. Henry, J. D., & Crawford, J. R. (2005). The short-form version of the Depression Anxiety Stress Scales (DASS-21): Construct validity and normative data in a large non-clinical sample. British journal of clinical psychology, 44(2), 227-239. https://doi.org/10.1348/014466505X29657
- [Background] 31. Hexel, M. (2004). Validierung der deutschen Version des Attachment Style Questionnaire (ASQ) bei Personen mit und ohne psychiatrische Diagnosen. Zeitschrift für Klinische Psychologie und Psychotherapie, 33(2), 79-90. Hogrefe Verlag. https://doi.org/10.1026/0084-5345.33.2.79
- [Background] 32. Hudecek, M. F. C., Blabst, N., Morgen, B., & Lermer, E. (2021). Eindimensionale Skala zur Messung von Dankbarkeit (GQ-5-G). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). https://doi.org./10.6102/zis300
- [Background] 33. Hughes, M. E., Waite, L. J., Hawkley, L. C., & Cacioppo, J. T. (2004). A short scale for measuring loneliness in large surveys: Results from two population-based studies. Research on aging, 26(6), 655-672. https://doi.org/10.1177/0164027504268574
- [Background] 34. Hupfeld, J., & Ruffieux, N. (2011). Validierung einer deutschen Version der Self-Compassion Scale (SCS-D). Zeitschrift Für Klinische Psychologie Und Psychotherapie, 40(2), 115-123. https://doi.org/10.1026/1616-3443/a000088
- [Background] 35. Kabat-Zinn, J. (1982). An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: Theoretical considerations and preliminary results. General hospital psychiatry, 4(1), 33-47. https://doi.org/10.1016/0163-8343(82)90026-3
- [Background] 36. Kabat-Zinn, J. (2003). Mindfulness-based interventions in context: Past, present, and future. Clinical Psychology: Science and Practice, 10(2), 144-156. https://doi.org/10.1093/clipsy.bpg016
- [Background] 37. Kinnunen, S. P., & Windmann, S. (2013). Inclusion of Other in Self Scale--German Version [Database record]. APA PsycTests. https://doi.org/10.1037/t62377-000
- [Background] 38. Kisley, M. A., Beblo, T., & Lac, A. (2025). Emotion Acceptance Questionnaire (EAQ): Factor Analysis and Psychometric Evaluation. Journal of Personality Assessment, 107(4), 516-529. https://doi.org/10.1080/00223891.2024.2444448
- [Background] 39. Klein, E. M., Brähler, E., Dreier, M. et al. (2016). The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry 16, 159 (2016). https://doi.org/10.1186/s12888-016-0875-9
- [Background] 40. Kliem, S., Mößle, T., Rehbein, F., Hellmann, D. F., Zenger, M., & Brähler, E. (2015). A brief form of the Perceived Social Support Questionnaire (F-SozU) was developed, validated, and standardized. Journal of clinical epidemiology, 68(5), 551-562. https://doi.org/10.1016/j.jclinepi.2014.11.003
- [Background] 41. Klimecki, O. M., Leiberg, S., Ricard, M., & Singer, T. (2014). Differential pattern of functional brain plasticity after compassion and empathy training. Social cognitive and affective neuroscience, 9(6), 873-879. https://doi.org/10.1093/scan/nst060
- [Background] 42. Knoll, N., Rieckmann, N., & Schwarzer, R. (2005). Coping as a mediator between personality and stress outcomes: a longitudinal study with cataract surgery patients. European Journal of Personality, 19(3), 229-247. https://doi.org/10.1002/per.546
- [Background] 43. Kok, B. E., & Singer, T. (2017a). Phenomenological fingerprints of four meditations: Differential state changes in affect, mind-wandering, meta-cognition, and interoception before and after daily practice across 9 months of training. Mindfulness, 8(1), 218-231. https://doi.org/10.1007/s12671-016-0594-9
- [Background] 44. Kok, B. E., & Singer, T. (2017b). Effects of contemplative dyads on engagement and perceived social connectedness over 9 months of mental training: A randomized clinical trial. JAMA Psychiatry, 74(2), 126-134. https://doi.org/10.1001/jamapsychiatry.2016.3360
- [Background] 45. Kroenke, K., Spitzer, R. L., & Williams, J. B. (2003). The Patient Health Questionnaire-2: validity of a two-item depression screener. Medical care, 41(11), 1284-1292. https://doi.org/10.1097/01.mlr.0000093487.78664.3c
- [Background] 46. Liedtke, C., Kohl, W., Kret, M. E., & Koelkebeck, K. (2018). Emotion recognition from faces with in-and out-group features in patients with depression. Journal of Affective Disorders, 227, 817-823. https://doi.org/10.1016/j.jad.2017.11.085
- [Background] 47. Loch, N., Hiller, W., & Witthöft, M. (2011). Der Cognitive Emotion Regulation Questionnaire (CERQ). Erste teststatistische Überprüfung einer deutschen Adaption [The Cognitive Emotion Regulation Questionnaire (CERQ). Psychometric evaluation of a German adaptation]. Zeitschrift für Klinische Psychologie und Psychotherapie: Forschung und Praxis, 40(2), 94-106. https://doi.org/10.1026/1616-3443/a000079
- [Background] 48. Löwe, B., Kroenke, K., Herzog, W., & Gräfe, K. (2004). Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). Journal of affective disorders, 81(1), 61-66. https://doi.org/10.1016/S0165-0327(03)00198-8
- [Background] 49. Löwe, B., Müller, S., Brähler, E., Kroenke, K., Albani, C., & Decker, O. (2007). Validierung und Normierung eines kurzen Selbstratinginstrumentes zur Generalisierten Angst (GAD-7) in einer repräsentativen Stichprobe der deutschen Allgemeinbevölkerung. PPmP-Psychotherapie Psychosomatik· Medizinische Psychologie, 57(02), A050.
- [Background] 50. Martin, A., Rief, W., Klaiberg, A., & Braehler, E. (2006). Validity of the brief patient health questionnaire mood scale (PHQ-9) in the general population. General hospital psychiatry, 28(1), 71-77. https://doi.org/10.1016/j.genhosppsych.2005.07.003
- [Background] 51. Maslach, C., & Jackson, S. E. (1981). The measurement of experienced burnout. Journal of organizational behavior 2(2), 99-113. https://doi.org/10.1002/job.4030020205
- [Background] 52. Matthäus, H., Heim, C., Voelke, M., Singer, T. (2024a). Reducing Neuroendocrine Psychosocial Stress Response Through Socio-emotional Dyadic but not Mindfulness Online Training. Frontiers in Endocrinology 15, 1277929. https://doi.org/10.3389/fendo.2024.1277929
- [Background] 53. Matthäus, H., Godara, M., Silveira, S. J., Hecht, M., Voelkle, M. C., Singer, T. (2024b). Loneliness through the Power of Practicing Together: A Randomized Controlled Trial of Online Dyadic Socio-Emotional vs. Mindfulness-Based Training. International Journal of Environmental Research and Public Health 21(5), 570. https://doi.org/10.3390/ijerph21050570
- [Background] 54. McCullough, M. E., Emmons, R. A., & Tsang, J.-A. (2002). The grateful disposition: A conceptual and empirical topography. Journal of Personality and Social Psychology, 82(1), 112-127. https://doi.org/10.1037/0022-3514.82.1.112
- [Background] 55. Moran, P., Leese, M., Lee, T., Walters, P., Thornicroft, G., & Mann, A. (2003). Standardised Assessment of Personality-Abbreviated Scale (SAPAS): preliminary validation of a brief screen for personality disorder. The British Journal of Psychiatry, 183(3), 228-232. https://doi.org/10.1192/bjp.183.3.228
- [Background] 56. Nilges, P. & Essau, C. (2021). DASS. Depressions-Angst-Stress-Skalen - deutschsprachige Kurzfassung [Verfahrensdokumentation und Fragebogen mit Auswertung]. In Leibniz-Institut für Psychologie (ZPID) (Hrsg.), Open Test Archive. Trier: ZPID. https://doi.org/10.23668/psycharchives.4579
- [Background] 57. Norris, J., Carpenter, J. G., Eaton, J., Guo, J. W., Lassche, M., Pett, M. A., & Blumenthal, D. K. (2015). The development and validation of the interprofessional attitudes scale: assessing the interprofessional attitudes of students in the health professions. Academic Medicine, 90(10), 1394-https://doi.org/10.1097/acm.0000000000000764
- [Background] 58. O'Malley, B., Linz, R., Engert, V., Singer, T. (2024). Testing the monitor and acceptance theory: the role of training-induced changes in monitoring-and acceptance-related capacities after attention-based, socio-emotional, or socio-cognitive mental training in reducing cortisol stress reactivity. Stress 27 (1), 2345906. https://doi.org/10.1080/10253890.2024.2345906
- [Background] 59. Paulus, C. M. (2009). Der Saarbrücker Persönlichkeitsfragebogen SPF(IRI) zur Messung von Empathie: Psychometrische Evaluation der deutschen Version des Interpersonal Reactivity Index. Saarbrücken: Universität des Saarlandes.
- [Background] 60. Peacock, E. J., & Wong, P. T. (1990). The stress appraisal measure (SAM): A multidimensional approach to cognitive appraisal. Stress medicine, 6(3), 227-236. https://doi.org/10.1002/smi.2460060308
- [Background] 61. Pedersen, T. H., Cignacco, E., Meuli, J., Habermann, F., Berger-Estilita, J., & Greif, R. (2020). The German interprofessional attitudes scale: Translation, cultural adaptation, and validation. GMS Journal for Medical Education, 37(3), Doc32. https://doi.org/10.3205/zma001325
- [Background] 62. Prendergast, M., Cardoso Pinto, A. M., Harvey, C. J., & Muir, E. (2024). Burnout in early year medical students: experiences, drivers and the perceived value of a reflection-based intervention. BMC Medical Education, 24(1), 7. https://doi.org/10.1186/s12909-023-04948-0
- [Background] 63. Qualter, P., Petersen, K., Barreto, M., Victor, C., Hammond, C., & Arshad, S. A. (2021). Exploring the frequency, intensity, and duration of loneliness: a latent class analysis of data from the BBC loneliness experiment. International Journal of Environmental Research and Public Health, 18(22), 12027. https://doi.org/10.3390/ijerph182212027
- [Background] 64. Raes, F., Pommier, E., Neff, K. D., & Van Gucht, D. (2011). Construction and factorial validation of a short form of the Self-Compassion Scale. Clinical Psychology & Psychotherapy, 18(3), 250-255. https://doi.org/10.1002/cpp.702
- [Background] 65. Ritz, T., & Kannapin, O. (2000). Zur Konstruktvalidität einer deutschen Fassung der Toronto Alexithymia Scale [The construct validity of a German version of the Toronto Alexithymia Scale]. Zeitschrift für Differentielle und Diagnostische Psychologie, 21(1), 49-64. https://doi.org/10.1024/0170-1789.21.1.49
- [Background] 66. Russell, D., Peplau, L. A., & Cutrona, C. E. (1980). The revised UCLA Loneliness Scale: Concurrent and discriminant validity evidence. Journal of Personality and Social Psychology, 39(3), 472-480. https://doi.org/10.1037/0022-3514.39.3.472
- [Background] 67. Russell, J. A., Weiss, A., & Mendelsohn, G. A. (1989). Affect grid: a single-item scale of pleasure and arousal. Journal of personality and social psychology, 57(3), 493. https://doi.org/10.1037/0022-3514.57.3.493
- [Background] 68. Sarubin, N., Gutt, D., Giegling, I., Bühner, M., Hilbert, S., Krähenmann, O., Wolf, M., Jobst, A., Sabaß, L., Rujescu, D., Falkai, P., & Padberg, F. (2015). Erste Analyse der psychometrischen Eigenschaften und Struktur der deutschsprachigen 10- und 25-Item Version der Connor-Davidson Resilience Scale (CD-RISC). European Journal of Health Psychology, 23(5). https://doi.org/10.1026/0943-8149/a000142
- [Background] 69. Silveira, S., Godara, M., & Singer, T. (2023). Boosting Empathy and Compassion Through Mindfulness-Based and Socioemotional Dyadic Practice: Randomized Controlled Trial With App-Delivered Trainings. Journal of Medical Internet Research, 25(1), e45027. https://doi.org/10.2196/45027
- [Background] 70. Sinclair, S., McClement, S., Raffin-Bouchal, S., Hack, T. F., Hagen, N. A., McConnell, S., & Chochinov, H. M. (2016). Compassion in health care: an empirical model. Journal of pain and symptom management, 51(2), 193-203. https://doi.org/10.1016/j.jpainsymman.2015.10.009
- [Background] 71. Singer, T. (2025). A neuroscience perspective on the plasticity of the social and relational brain. Annals of the New York Academy of Sciences, 1547(1), 52-74. https://doi.org/10.1111/nyas.15319
- [Background] 72. Singer, T., & Engert, V. (2019). It matters what you practice: Differential training effects on subjective experience, behavior, brain and body in the ReSource Project. Current Opinion in Psychology, 28, 151-158. https://doi.org/10.1016/j.copsyc.2018.12.005
- [Background] 73. Singer, T. & Klimecki, O. (2014). Empathy and compassion. Current Biology 24 (18), S. R875 - R878. https://doi.org/10.1016/j.cub.2014.06.054
- [Background] 74. Singer, T., Kok, B. E., Bornemann, B., Bolz, M., & Bochow, C. (2015). The ReSource Project: Background, design, samples, and measurements (1st ed.). Leipzig: Max Planck Institute for Human Cognitive and Brain Sciences. https://hdl.handle.net/21.11116/0000-0003-FEC8-E
- [Background] 75. Söchtig, A., Kliem, S., & Kröger, C. (2012). Diagnostik Efficiency of the German Version of the Self-Rated Standardized Assessment of Personality-Abbreviated Scale. Psychopathology, 45(6), 381 - 389. https://doi.org/10.1159/000337970
- [Background] 76. Spitzer, R. L., Kroenke, K., Williams, J. B., & Lowe, B. (2006). A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of Internal Medicine, 166(10),1092-1097. https://doi.org/10.1001/archinte.166.10.1092
- [Background] 77. Teasdale, J. D., Segal, Z. V., Williams, J. M. G., Ridgeway, V. A., Soulsby, J. M., & Lau, M. A. (2000). Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. Journal of Consulting and Clinical Psychology, 68(4), 615-623. https://doi.org/10.1037/0022-006X.68.4.615
- [Background] 78. Wang, Z., Wu, P., Hou, Y. Guo, J., & Lin, C. (2024) The effects of mindfulness-based interventions on alleviating academic burnout in medical students: a systematic review and meta-analysis. BMC Public Health 24, 1414. https://doi.org/10.1186/s12889-024-18938-4